CLINICAL TRIAL: NCT00339170
Title: Cognitive Training and Enhanced Supported Employment
Brief Title: Cognitive Training and Enhanced Supported Employment in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH061493 (NIH); R01MH061493 (NIH); DSIR AT-RH
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder; Schizophrenic Disorders; Psychotic Disorders; Cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants receive a 12-month cognitive enhancement training program plus a 12-month work therapy program.
  Interventions: Behavioral: Computer-Based Cognitive Enhancement Training Program; Behavioral: Work Therapy Program
- 2 (Active Comparator): Participants receive a 12-month work therapy program alone.
  Interventions: Behavioral: Work Therapy Program

INTERVENTIONS:
Behavioral: Computer-Based Cognitive Enhancement Training Program — Participants in the cognitive enhancement training program will receive feedback on their cognitive strengths and weaknesses based on the outcomes of the baseline assessment. The training component will be comprised of 150 computer-based exercises that focus on improving memory, attention, and organizational skills. Participants will attend two weekly meetings: one will focus on providing feedback regarding goal-setting and problem-solving, and the other will focus on improving verbal skills and social information processing.
  Arms: 1
Behavioral: Work Therapy Program — Participants in the work therapy program will attend two non-cognitive discussion groups per week.

SUMMARY:
This study will evaluate the effectiveness of a computer-based cognitive enhancement program plus a work therapy program at improving productivity, work performance, and quality of life in schizophrenic individuals.

DETAILED DESCRIPTION:
Schizophrenia is a chronic, severe, and disabling brain disorder that affects 2.4 million people in the United States. Individuals with schizophrenia may have difficulties with cognitive functioning, including problems with attention, memory, and organizational thought processes. These factors can lead to decreased productivity and poor work performance, which may make holding a job difficult. Research has shown that certain types of psychological therapies, such as cognitive behavioral therapy, are useful in reducing the severity of schizophrenic symptoms. The purpose of this study is to determine whether a computer-based cognitive enhancement training program, in combination with a work therapy program, will enhance workplace performance, productivity, and quality of life in individuals with schizophrenia.

This study will enroll individuals with schizophrenia or schizoaffective disorder. Participants will undergo a cognitive assessment at baseline. They will then be randomly assigned to either a 12-month cognitive enhancement training program plus a 12-month work therapy program or a 12-month work therapy program alone. Participants in the cognitive enhancement training program will receive feedback on their cognitive strengths and weaknesses based on the outcomes of the baseline assessment. The training component will be comprised of 150 computer-based exercises that focus on improving memory, attention, and organizational skills. Participants will attend two weekly meetings: one will focus on providing feedback regarding goal-setting and problem-solving, and the other will focus on improving verbal skills and social information processing. Individuals taking part only in the work therapy program will attend two non-cognitive discussion groups per week. All participants will work up to 20 hours a week in an approved work environment, and will have access to appropriate support services. Following the end of the program, participants will have the option of working an additional 12 months. Schizophrenia symptoms, quality of life, and neuropsychological and rehabilitation effects will be assessed at the end of Years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* Hospitalized in the 30 days prior to study entry
* Homeless in the 30 days prior to study entry
* Changed medications in the 30 days prior to study entry
* Substance abuse in the 30 days prior to study entry
* History of head trauma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2000-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Schizophrenia symptoms | Measured at Year 1
Vocational functioning | Measured at Year 2
Schizophrenia symptoms | Measured at Year 2
Quality of life | Measured at Year 2
Quality of life | Measured at Year 1
Vocational functioning | Measured at Year 1

SECONDARY OUTCOMES:
Number of hospitalizations | Measured at Year 1
Income | Measured at Year 1
Number of hospitalizations | Measured at Year 2
Income | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Bell, PhD, Principal Investigator — Yale University School of Medicine, VA CT Healthcare System
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Bell, M.D., Bryson, G., Kaplan, E. Work rehabilitation in schizophrenia: cognitive predictors of best and worst performance. Schizophrenia Research. 1999; 36:322.
- [Background] Bell M, Bryson G, Wexler BE. Cognitive remediation of working memory deficits: durability of training effects in severely impaired and less severely impaired schizophrenia. Acta Psychiatr Scand. 2003 Aug;108(2):101-9. doi: 10.1034/j.1600-0447.2003.00090.x. PMID 12823166
- [Background] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Background] Bell MD, Fiszdon J, Bryson G, Wexler BE. Effects of neurocognitive enhancement therapy in schizophrenia: normalisation of memory performance. Cogn Neuropsychiatry. 2004 Aug;9(3):199-211. doi: 10.1080/13546800344000084. PMID 16571581
- [Background] Greig T, Zito W, Bell MD. Rehab rounds: A hybrid transitional and supported employment program. Psychiatr Serv. 2004 Mar;55(3):240-2. doi: 10.1176/appi.ps.55.3.240. No abstract available. PMID 15001722
- [Background] Bell, M.D., Brsyon, G.J. Work rehabilitation in schizophrenia: cognitive predictors of best and worst performance. Schizophrenia Research. 2001;36:322.
- [Background] Bell, M.D, Brsyon, G.J , Fiszdon, J., Greig, T.C., Wexler, B.E. Neurocognitive enhancement therapy and work therapy in schizophrenia: Work outcomes at 6 months and 12 month follow-up. Biological Psychiatry. 2004; 55: 1S-242S.
- [Background] Greig, T.C., Nicholls, S.S., Bryson, G.J., Bell, M.D. The Vocational Cognitive Rating Scale: A Scale for the Assessment of Cognitive Functioning at Work for Clients With Severe Mental Illness. The Journal of Vocational Rehabilitation. 2004; 21: 71-81.
- [Background] Bryson, G & Bell, MD. Work performance improvement in schizophrenia: Symptom and cognitive predictors. Schizophrenia Resarch. 2001; 49: 258.
- [Derived] Bell MD, Choi KH, Dyer C, Wexler BE. Benefits of cognitive remediation and supported employment for schizophrenia patients with poor community functioning. Psychiatr Serv. 2014 Apr 1;65(4):469-75. doi: 10.1176/appi.ps.201200505. PMID 24382594
- [Derived] Surti TS, Corbera S, Bell MD, Wexler BE. Successful computer-based visual training specifically predicts visual memory enhancement over verbal memory improvement in schizophrenia. Schizophr Res. 2011 Nov;132(2-3):131-4. doi: 10.1016/j.schres.2011.06.031. Epub 2011 Jul 27. PMID 21795025